CLINICAL TRIAL: NCT05009212
Title: Randomized Trial of Endoscopic Stricturotomy Versus Endoscopic Balloon Dilatation in Patients With Crohn's Disease and Symptomatic Small Bowel Stricture
Brief Title: Endoscopic Stricturotomy Versus Endoscopic Balloon Dilatation in Patients With Crohn's Disease and Symptomatic Small Bowel Stricture
Acronym: DESTRESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021ZSLYEC-243
Record Dates: First submitted 2021-08-08; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Crohn Disease; Stricture; Bowel; Endoscopy, Gastrointestinal
MeSH Terms: conditions — Crohn Disease; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESt group (Experimental): Endoscopic stricturotomy
  Interventions: Procedure: Endoscopic stricturotomy
- EBD group (Active Comparator): Endoscopic balloon dilatation
  Interventions: Procedure: Endoscopic balloon dilatation

INTERVENTIONS:
Procedure: Endoscopic stricturotomy — Endoscopic stricturotomy for bowel stricture (<5 cm)
  Arms: ESt group
Procedure: Endoscopic balloon dilatation — Endoscopic balloon dilatation for bowel stricture (<5 cm)
  Arms: EBD group

SUMMARY:
Stenosis is one of the most frequent complications in patients with Crohn's disease (CD). In particular, CD patients with intestinal strictures are often faced with short bowel syndrome after repeated or extensive surgical resection.

Endoscopic management shows good efficacy and safety in the treatment of strictures in CD patients. The European Crohn's and Colitis Organisation (ECCO) guideline recommended that endoscopic balloon dilatation is suitable to treat short [<5 cm] strictures of the terminal ileum in CD. Recently, Lan et al. reported that endoscopic stricturotomy appeared to be more effective in treating CD patients with anastomotic stricture than endoscopic balloon dilatation.

However, there is no prospective clinical studies evaluating the efficacy and safety of endoscopic stricturotomy in the treatment of fibrostenotic Crohn's disease. The trial aims to compare the efficacy and safety of endoscopic stricturotomy with endoscopic balloon dilation in the treatment of small bowel stricture in patients with Crohn's Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects had been diagnosed with CD for at least 3 months prior to screening, and the diagnosis of CD had clinical findings and endoscopic, imaging evidence, and was supported by histopathology reports
2. Subject is in remission from CD (CDAI score < 150)
3. Subjects had clinical findings of multiple fibrotic strictures of the bowel with obstruction and imaging evidence, and/or endoscopic evidence
4. Subjects had ≤ 3 small bowel strictures (length < 5 cm) from duodenum to rectum and < 50 cm distance between strictures
5. Study process prior to initiation, the subject or subject's legal representative (if applicable) signed and dated a written informed consent form or any required documentation of privacy authorization
6. Female subjects who remained sexually and of childbearing potential with an ungerminated male partner, consented to adequate routine contraception throughout the study period starting with signing informed consent

Exclusion Criteria:

1. At the initial screening visit, subject presented with enterocutaneous fistula, abdominal abscess, evidence of gastrointestinal bleeding
2. Subjects were in active CD (CDAI score ≥ 150)
3. The subject had inflammatory activity in the stenotic bowel (as judged by a combination of blood inflammatory indices, endoscopy, ultrasound and imaging)
4. Presence of ileostomy, colostomy
5. Subjects had a history or evidence of adenomatous colonic polyps that had not been resected or had a history or evidence of dysplasia of the colonic mucosa, including low - or high-grade dysplasia, and an undiagnosed type of dysplasia
6. Subjects had suspected or confirmed ulcerative colitis, undiagnosed types of colitis, ischemic colitis, radiation enteritis, colitis associated diverticular disease, or microscopic colitis
7. Subjects had evidence of active infection during the screening period
8. Subject has active tuberculosis
9. Subjects with any defined inborn or acquired immunodeficiency (e.g., common various immunodeficiencies, human immunodeficiency virus [HIV] infection, organ transplantation)
10. Subjects had a clinically significant infection (e.g., pneumonia, pyelonephritis) or an ongoing chronic infection within 30 days prior to screening
11. The subject suffered from any unstable or uncontrolled cardiovascular, pulmonary, hepatic, renal, gastrointestinal, genitourinary, hematological, coagulation, immune, endocrine / metabolic or other medical condition that, in the opinion of the investigator, would interfere with the outcome of the study or jeopardize the safety of the subject
12. The subject's medical history included malignancy
13. Subjects had abnormal laboratory results for any of the following during screening: hemoglobin < 5 g / dl; white blood cell (WBC) count < 3 ×10E9 / L; platelet count < 100 × 10E9 / L or > 1200 × 10E9 / L; alanine transaminase (ALT) or aspartate transaminase (AST) > 3 × upper limit of normal (ULN), and serum creatinine > 2 × ULN.
14. Subjects were unable to attend all study visits or comply with study flow plans female subjects were pregnant prior to study enrollment, during study enrollment, or plan to donate eggs during these time periods
15. Subjects were forced to consent to participate in the study
16. Investigators considered the subject unsuitable for endoscopic treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Surgery-free survival | 52 weeks
  Percentage of patients who do not receive surgical intervention for obstruction recurrence

SECONDARY OUTCOMES:
Endoscopic intervention-free survival | 52 weeks
  Percentage of patients who do not receive endoscopic intervention for obstruction recurrence
Intervention-free survival | Week 52
  Percentage of patients who do not receive surgical or endoscopic intervention for obstruction recurrence
Technical success rate | Week 0
  The passage of endoscope without resistance
Obstructive score change | Week 8, 16, 26, 52
  Obstructive score (scaling from 0 to 6, higher scores mean a worse outcome) change compared to baseline
Crohn's Disease Activity Index (CDAI) score change | Week 8, 16, 26, 52
  Higher scores mean a worse outcome for CDAI score
Inflammatory Bowel Disease Questionnaire (IBDQ) score reduction | Week 8, 16, 26, 52
  Higher scores mean a better outcome for IBDQ score
Adverse event rate | Week 52
  Percentage of adverse events
Total cost | Week 52
  Total cost for intervention

CONTACTS AND LOCATIONS:
Overall Officials: Qin Guo, MD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No